CLINICAL TRIAL: NCT06791590
Title: Evaluating the Effects of Intermittent Oro-esophageal in Tracheotomy Patients With Neurogenic Dysphagia: a Randomized Study
Brief Title: Evaluating the Effects of Intermittent Oro-esophageal in Tracheotomy Patients With Neurogenic Dysphagia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jingyi Ge, Principal Investigator, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025bkky-003
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Neurogenic Dysphagia; Tracheotomy Patients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): Intranasal continuous nasogastric tube or nasogastric tube nutritional support was used. For patients at risk of repeated aspiration and regurgitation, patients with gastric nutritional intolerance who could not be improved by using gastrointestinal motility drugs, intestinal indentation tube and retropyloric feeding were given.
  Interventions: Procedure: Naso-intestinal tube nutrition support
- experimental group (Experimental): Disposable gastric tube was used for enteral nutrition support
  Interventions: Procedure: intermittent oro-esophageal

INTERVENTIONS:
Procedure: intermittent oro-esophageal — A disposable gastric tube was used to perform enteral nutrition support therapy, and contraindications were evaluated again. Inform the patient and family members of the precautions for intermittent feeding through oral tube, and play the video of the operation process to make them actively cooperate with the operation.
  Arms: experimental group
Procedure: Naso-intestinal tube nutrition support — For patients at risk of repeated aspiration and regurgitation, and for patients with gastric nutritional intolerance that cannot be improved by gastrointestinal motivity drugs, indwelling intestinal tube and retropyloric feeding are given.
  Arms: Control group

SUMMARY:
Neurogenic dysphagia refers to swallowing disorders caused by the damage of swallowing central or peripheral nerves and muscles. According to statistics, about 50% of patients with neurological diseases will be complicated with neurogenic dysphagia. Common diseases include stroke, dementia, Parkinson's disease and neuromuscular diseases. Dysphagia has a great impact on the quality of life of patients, and is related to malnutrition, aspiration pneumonia and even death. In severe cases, tracheotomy is required to maintain airway patency and discharge secretions. The common nutritional support methods for patients with neurogenic dysphagia after tracheotomy are nasogastric or nasointestinal tube placement and percutaneous gastrostomy.

intermittent oro-esophageal tube feeding (IOE) is a new nutrition method proposed by scholars in recent years. Studies have shown that it can improve the swallowing function of patients with dysphagia while meeting the nutritional needs of patients, so as to effectively improve the quality of life of patients. However, there are few studies on patients with dysphagia after tracheotomy. This study aims to compare the intervention effects of two kinds of tube feeding methods in patients with neurogenic dysphagia after tracheotomy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of neurogenic dysphagia；
* Acute phase has passed, weaning time > 48 hours, tracheotomy time >1 week; in accordance with the decannulation process of tracheotomy patients formulated by our center in 2018;
* steady vital signs, without severe cognitive impairment or sensory aphasia, able to cooperate with the assessment；
* Gastrointestinal motility is good, can tolerate more than 150ml/h feeding pump speed;
* Willing to sign an informed consent form.

Exclusion Criteria:

* Structural swallowing disorders, such as oral, pharyngeal, larynx, esophagus and other anatomical abnormalities caused by swallowing disorders;
* The clinical condition was unstable, accompanied by heart, lung, brain and other important organ dysfunction;
* Severe cognitive dysfunction, confusion, unable to cooperate.

Ages: 18 Years to 92 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-01-28 (Estimated); Primary Completion 2025-02-10 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Decannulation time of the tracheostomy tube | 6 month

SECONDARY OUTCOMES:
Decannulation rate | 6 month
Flexible endoscopic examination of swallowing | 6 month
Nutritional status-albumin | 6 month
Swallowing Quality of Life questionnaire | 6 month
leakage-aspiration grade | 6 month